CLINICAL TRIAL: NCT05828589
Title: A Phase 1/1b Open-Label Dose-Escalation and Dose-Optimization Study of Bcl-2 Inhibitor BGB-21447 in Patients With Mature B-Cell Malignancies
Brief Title: A Study of BGB-21447, a Bcl-2 Inhibitor, in Mature B-Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-21447-101; CT-2023-CTN-05421-1 (Other: Australia Clinical Trial Number); CTR20231287 (Other: ChinaDrugTrials); 2025-521600-21-00 (EU CTIS Number)
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Relapsed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Relapsed Follicular Lymphoma; Relapsed Marginal Zone Lymphoma; Relapse Diffuse Large B Cell Lymphoma; Relapsed Small Lymphocytic Lymphoma; Refractory Follicular Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Small Lymphocytic Lymphoma; Richter Transformation; Refractory Diffuse Large B-cell Lymphoma; Transformed Non-Hodgkin Lymphoma
Keywords: Relapsed Non-Hodgkin Lymphoma; refractory non-Hodgkin lymphoma; Relapsed Chronic Lymphocytic Leukemia; Follicular Lymphoma; Marginal Zone Lymphoma; NHL; FL; MZL; Refractory Chronic Lymphocytic Leukemia; RCLL; Relapsed Follicular Lymphoma; Refractory Follicular Lymphoma; Relapsed Marginal Zone Lymphoma; Refractory Marginal Zone Lymphoma; RFL; RMZL; Relapsed Small Lymphocytic Lymphoma; Refractory Small Lymphocytic Lymphoma; RSLL; Richter's transformation; RT; RR DLBCL; Bcl-2; Bcl-2i
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Cohort A1): Dose escalation in patients with B-cell non-Hodgkin lymphoma (NHL) (Experimental): Participants with R/R B-cell NHL (including diffuse large B-cell lymphoma [DLBCL], follicular lymphoma [FL], marginal zone lymphoma [MZL], transformed B-cell NHL (B-NHL), and Richter's transformation to DLBCL) will receive BGB-21447 once a day.
  Interventions: Drug: BGB-21447
- Part 1 (Cohort B): Dose escalation in R/R CLL/SLL participants with low tumor burden (Experimental): Participants with relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) will receive BGB-21447 once a day.
  Interventions: Drug: BGB-21447
- Part 2 (Cohort A2.1): BGB-21447 Monotherapy Dose Optimization in R/R DLBCL (Experimental): Participants will receive BGB-21447 with two dose levels from Cohort A1 for further evaluation of safety and efficacy.
  Interventions: Drug: BGB-21447
- Part 2 (Cohort A2.2): BGB-21447 Monotherapy Dose Optimization in R/R FL or R/R MZL (Experimental): Participants will receive BGB-21447 with two dose levels from Cohort A1 for further evaluation of safety and efficacy.
  Interventions: Drug: BGB-21447

INTERVENTIONS:
Drug: BGB-21447 — BGB-21447 will be administered orally

SUMMARY:
This study is testing the safety and tolerability of BGB-21447 monotherapy in participants with relapsed or refractory (R/R) non-Hodgkin lymphoma (NHL) and chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL). The study aims to determine the maximum tolerated dose (MTD), maximum administered dose (MAD), recommended Phase 2 dose (RP2D), and pharmacokinetic profile of the drug. Additionally, preliminary antitumor activity will be characterized. The study is divided into 2 main parts: Part 1 "Monotherapy Dose Finding" and Part 2 "Monotherapy Dose Optimization."

ELIGIBILITY:
Inclusion Criteria

1. Confirmed diagnosis (per World Health Organization [WHO] guidelines, unless otherwise noted) of one of the following:

   Cohort A1 and Cohort A2:
   1. R/R DLBCL (for Cohort A1 and Cohort A2.1)

      * High-grade B-cell lymphomas with translocations of MYC and Bcl-2 and/or Bcl-6 are not allowed in Cohort A1 but may be allowed in Cohort A2.1
   2. R/R FL (for Cohort A1 and Cohort A2.2)
   3. R/R MZL (for Cohort A1 and Cohort A2.2)
   4. Transformed B-cell NHL (for Cohort A1 only)
   5. Richter's transformation to DLBCL (for Cohort A1 only)
2. Measurable disease by computed tomography/magnetic resonance imaging.

Exclusion Criteria:

1. Prior malignancy (other than the disease under study) within the past 2 years, except for curatively treated basal or squamous skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score ≤ 6 prostate cancer or lentigo maligna melanoma that has been curatively resected
2. Known central nervous system involvement by lymphoma/leukemia
3. Prior autologous stem cell transplant < 3 months before the first dose of study drug. Or prior chimeric antigen receptor T-cell (CAR-T) therapy < 3 months before the first dose of study drug
4. Prior allogeneic stem cell transplant.
5. Major surgery < 4 weeks before the first dose of study treatment

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose limiting toxicities (DLTs) | Up to approximately 1 month
  Number of participants with dose limiting toxicities, as defined in the study protocol.
Number of participants with adverse events (AEs) | From the first dose of study drug to 30 days after the last dose or initiation of new anticancer therapy, whichever occurs first; up to approximately 12 months
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) assessed and graded based upon the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0).
Number of participants with Tumor Lysis Syndrome (TLS) | From the first dose of study drug to 30 days after the last dose or initiation of new anticancer therapy, whichever occurs first; up to approximately 12 months
  TLS will be determined via laboratory values and assessed by the investigator.
  In laboratory tumor lysis syndrome, 2 or more metabolic abnormalities must be present during the 24-hour period within 3 days before the start of study drug treatment or up to 7 days afterward. Clinical tumor lysis syndrome requires the presence of laboratory tumor lysis syndrome plus an increased creatinine level, seizures, cardiac dysrhythmia, or death.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) After a Single Dose of BGB-21447 | Up to approximately 8 weeks
Area under the curve from time 0 to the last sampling time point within the dose interval (AUC0-t) After a Single Dose of BGB-21447 | Up to approximately 8 weeks
Area under the curve from time 0 extrapolated to infinity time (AUCinf) After a Single Dose of BGB-21447 | Up to approximately 8 weeks
Time to reach maximum observed plasma concentration (Tmax) After a Single Dose of BGB-21447 | Up to approximately 8 weeks
Apparent terminal elimination half-life (t1/2) After a Single Dose of BGB-21447 | Up to approximately 8 weeks
Apparent oral clearance (CL/F) After a Single Dose of BGB-21447 | Up to approximately 8 weeks
Apparent volume of distribution (Vz/F) After a Single Dose of BGB-21447 | Up to approximately 8 weeks
Steady state maximum observed plasma concentration (Cmax,ss) of BGB-21447 | Up to approximately 8 weeks
Steady state pre-dose trough concentration (Ctrough,ss) of BGB-21447 | Up to approximately 8 weeks
Steady state area under the curve from time 0 to the quantifiable concentration (AUClast,ss) of BGB-21447 | Up to approximately 8 weeks
Steady state time to reach maximum observed plasma concentration (Tmax,ss) of BGB-21447 | Up to approximately 8 weeks
Overall response rate (ORR) | Up to approximately 24 months
  Defined as the percentage of patients who achieve partial response or better for diffuse large B-cell lymphoma, marginal zone lymphoma, follicular lymphoma, transformed B-NHL, and Richter's transformation to DLBCL as per the Lugano Classification for non-Hodgkin lymphoma.
Duration of Response (DOR) | Up to approximately 24 months
  Defined as the time from the first response documentation to the date that progression is documented after treatment initiation or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to approximately 24 months
  Defined as the time from treatment initiation to the first documentation of response.
Progression-free survival (PFS) | Up to approximately 24 months
  Defined as the time from treatment initiation to the first documented disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (28):
- United States (7):
  - Sibley Memorial Hospital Johns Hopkins Medicine, Washington D.C., District of Columbia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mission Cancer and Blood, Waukee, Iowa
  - Sidney Kimmel Comprehensive Cancer At Johns Hopkins, Baltimore, Maryland
  - Nyu Langone Health Perlmutter Cancer Center At Nyu Langone Hospital Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center At Nyu Langone Health, New York, New York
  - Avera Cancer Institute, Sioux Falls, South Dakota
- Australia (5):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (15):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central Peoples Hospitaljiangnan Branch, Yichang, Hubei
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University Branch Xianghu, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Linyi Peoples Hospital, Linyi, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/